CLINICAL TRIAL: NCT00060086
Title: Phase II Study Evaluating Pomegranate Juice In Patients With Recurrent Adenocarcinoma Of The Prostate
Brief Title: Pomegranate Juice in Treating Patients With Recurrent Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: POM Wonderful LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-001265; UCLA-0210049; CDR0000299439 (Other: UCLA IRB)
Record Dates: First submitted 2003-05-06; First posted 2003-05-07 (Estimated); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pomegranate Juice (Experimental): Subjects are given oral pomegranate juice once daily. Treatment continues for 18 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Dietary Supplement: pomegranate juice

INTERVENTIONS:
Dietary Supplement: pomegranate juice — Subjects receive oral pomegranate juice once daily. Treatment continues for 18 months in the absence of disease progression or unacceptable toxicity.

SUMMARY:
RATIONALE: Pomegranate juice may contain substances that decrease or slow the rise of prostate-specific antigen (PSA) levels and may be effective in delaying or preventing recurrent prostate cancer.

PURPOSE: This phase II trial is studying how well pomegranate juice works in decreasing or slowing the rise of PSA levels in patients who have undergone radiation therapy or surgery for prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether pomegranate juice can decrease or slow rising prostate-specific antigen (PSA) levels in patients who have undergone radical prostatectomy or radiotherapy for adenocarcinoma of the prostate.

OUTLINE: Patients receive oral pomegranate juice once daily. Treatment continues for 18 months in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 29-40 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate
* Must have undergone prior surgery or radiotherapy for the primary tumor
* Documented rising prostate-specific antigen (PSA) level, defined by the following criteria:
* Absolute level of PSA at least 0.2 ng/mL but less than 5.0 ng/mL
* Rising PSA level must be confirmed at least 1 week later
* Adequate PSA time points to calculate a PSA doubling time
* Gleason score no greater than 7
* Age 18 and over
* Performance status ECOG 0-1
* Life expectancy at least 6 months
* No other malignancy within the past 5 years except nonmelanoma skin cancer
* No other serious concurrent systemic medical disorders that would preclude study compliance
* No known allergy to pomegranate juice
* More than 4 weeks since prior participation in another experimental study

Exclusion Criteria:

* nodal involvement
* evidence of metastatic disease
* prior hormonal therapy
* concurrent hormonal therapy for rising PSA levels after initial therapy for prostate cancer
* concurrent participation in another experimental study
* other concurrent systemic or local therapy for prostate cancer
* initiation or discontinuation of any new nutritional or dietary supplements during study participation

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2004-11-30 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2021-05-25 (Actual)

PRIMARY OUTCOMES:
Clinical efficacy, in terms of overall response rate, measured by serum prostate-specific antigen (PSA) levels every 3 months | Evaluated every 3 months for 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Allan Pantuck, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States